CLINICAL TRIAL: NCT02687971
Title: A Randomized, Open Label, Multicenter Study to Determine the Efficacy and Safety of Combining Thermotherapy and a Short Course of Miltefosine for the Treatment of Uncomplicated Cutaneous Leishmaniasis in the New World¨
Brief Title: Thermotherapy + a Short Course of Miltefosine for the Treatment of Uncomplicated Cutaneous Leishmaniasis in the New World¨
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-MILT-07-CL
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermotherapy alone (Active Comparator): Local heat will be applied using a Localized Current Field radio-frequency generating device manufactured by Thermo-Med Technologies, Inc. A wand with 2 electrodes is connected to the main housing by a thin wire. The electrodes are applied to the skin. We will use electrodes 6 mm long, separated by 4 mm. One single session at the site of the lesion(s) at 50°C for 30" applications will be used. Depending on the size of the lesion, more than one application may be administered.
  Interventions: Drug: Miltefosine
- Thermotherapy plus Miltefosine (Experimental): In addition to receiving one single session of thermotherapy as described above, subjects will receive oral miltefosine two or three capsules a day, which is the equivalent of 100 to 150mg respectively for 21 days. Miltefosine capsules will be taken after breakfast, lunch and dinner, in other words, after food.
  The daily dose of miltefosine will depend on the weight of each patient. According to dosage instructions if the patient is taking the miltefosine twice a day, it must be taken in the morning and night (dose of 100mg/Kg/day). Whereas if the patient is taking miltefosine three times a day, it must be taken in the morning, noon and night (dose of 150mg/Kg/day).
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — Miltefosine (hexadecylphosphocholine) is an oral drug which has proven to be effective for the treatment of Visceral leishmaniasis (VL) in the Indian sub-continent. It has also been tested for CL, yielding varying results. Miltefosine was approved by FDA in 2014 for the treatment of CL in the New World for lesions due to L. braziliensis, L. panamensis and L. guyanensis only.
  Other Names: Impavido

SUMMARY:
The purpose of this trial is to determine the efficacy and safety of a combined therapy using thermotherapy (TT) (one session, 50 degrees Celsius for 30") + miltefosine at a standard dose of 2.5 mg/kg/day for 21 days for the treatment of uncomplicated CL in Peru and Colombia

DETAILED DESCRIPTION:
The use of topical treatments for Cutaneous leishmaniasis (CL) is an option that has been widely explored and it is currently listed as an options by WHO in those situations where the patient has few lesions (≤ 4) of less than ≤ 4 cm in diameter and located in areas of the body which may be treated topically.

Local heat, especially the one produced by radio frequency waves (Themo-Med®) has been widely tested for CL in both Old and New World. The advantages of using thermotherapy include: 1) high security profile; 2) only one session is required which ensures compliance with treatment; 3) easy to use in the field since the machine operates with batteries; 4) its effectiveness does not depend on the species of Leishmania causing the lesion as it is a physical measure; and 5) it can be used in patients in whom systemic treatment with antimonials are contraindicated, including women who are pregnant or breastfeeding. In the New World, Thermo-Med® has been evaluated in Mexico, Guatemala, Colombia and Brazil (all but one were randomized clinical trials), reporting cure rates of 90%, 73%, 64% and 75% respectively

There are no clinical trials evaluating the efficacy of miltefosine for CL when given for less than 20 days. The 21-day course was chosen to give the best chances to the combination approach and based on a) the results of a Phase II trial conducted in Colombia showing that a mean dose of miltefosine of 133 mg/day/20 days resulted in a cure rate of 82%20 and; b) a report showing that the a daily administration of 100 mg/day (2.5 mg/kg of body weight/day for 28 days) resulted in a mean maximum concentration of drug in serum at day 23 of treatment of 70,000 ng/ml21.

The theoretical advantages offered by this combination are that a) we are using two approaches that are currently recommended for use individually and for which there is good information regarding their efficacy and safety when used alone; b) the use of a topical plus a systemic treatment would hypothetically have an additive effect, since systemic treatment would eliminate those circulating or remaining parasites located in the periphery of the lesion that topical treatment fails to remove and which might be the cause of relapses22,23; c) it offers the opportunity to increase the current cure rate reported with any other treatment approach available when used alone; d) it will reduce the length of treatment with miltefosine and hopefully the cost and rates of adverse events associated with 28 days of treatment with miltefosine.

ELIGIBILITY:
Inclusion Criteria:

Patient with a confirmed diagnosis of CL in at least one lesion by at least one of the following methods: 1) microscopic identification of amastigotes in stained lesion tissue, or 2) demonstration of Leishmania by PCR, or 3) positive culture for promastigotes,

Patient has a lesion that satisfies the following criteria:

* Lesion size ≥ 0.5 cm and </= 4 cm (Longest diameter),
* Not located on the ear, face, close to mucosal membranes, joints or on a location that in the opinion of the PI is difficult to apply TT,
* Patient with </= 4 CL lesions,
* Duration of lesion less than 4 months by patient history, Patient able to give written informed consent, In the opinion of the investigator, the patient is capable of understanding and complying with the protocol

Exclusion Criteria:

* Female with a positive urine pregnancy test at screening or who is breast feeding, lactating or female at fertile age who does not agree to take appropriate contraception during treatment period and up to D90,
* History of clinically significant medical problems / treatment that might interact, either negatively or positively, with topical treatment of leishmaniasis including any immunocompromising condition,
* Within 8 weeks (56 days) of trial Day 1, received treatment for leishmaniasis with any medication including antimonials likely, in the opinion of the PI, to modify the course of the Leishmania infection,
* Has diagnosis or suspected diagnosis of mucocutaneous leishmaniasis based on physical exam,
* History of known or suspected hypersensitivity or idiosyncratic reactions to trial medication or exipients,
* Patient who is not willing to attend the trial visits, or is not able to comply with follow-up visits up to 6 months,
* Known history of drug addiction and/or alcohol abuse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Initial cure rate | Day 90, after start of treatment
  Initial Cure: Ulcerated lesions: 100% re-epithelialization of the lesion(s) by Day 90.
  Non-Ulcerated lesions: flattening and/or no signs of induration of the lesion(s) by Day 90.
  The percentage of re-epithelialization of the lesion(s) is calculated by comparing the size of the ulcer at Day 7 against the size at the follow up visit

SECONDARY OUTCOMES:
Final cure rate | Day 180, after star of treatment
  The number of patients who fulfill the criteria of initial cure and have no relapse by Day 180
Frequency and severity of AEs | Day 45
  Frequency and severity of AEs by treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Dario Velez, Prof, Principal Investigator — PECET, Universidad de Antioquia, Medellin, Colombia; Alejandro Llanos-Cuentas, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia, Lima, Peru
Locations (2):
- Programa de Estudios y Control de Enfermedades Tropicales (PECET), Universidad de Antioquia, Medellín, Colombia
- IMT Alexander Von Humboldt, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez L, Valencia B, Alvarez F, Ramos AP, Llanos-Cuentas A, Echevarria J, Velez I, Boni M, Rode J, Quintero J, Jimenez A, Tabares Y, Mendez C, Arana B. A phase II multicenter randomized study to evaluate the safety and efficacy of combining thermotherapy and a short course of miltefosine for the treatment of uncomplicated cutaneous leishmaniasis in the New World. PLoS Negl Trop Dis. 2022 Mar 7;16(3):e0010238. doi: 10.1371/journal.pntd.0010238. eCollection 2022 Mar. PMID 35255096